CLINICAL TRIAL: NCT03727191
Title: Evaluation of the Effect of the Consumption of a Hypercaloric/Hyperproteic Formula in the Coverage of Nutritional Requirements in Patients With Chewing/Swallowing Problems That Require a Shredded Diet.
Brief Title: Coverage of Requirements After Consumption of a Nutritional Formula in Patients With Chewing/Swallowing Problems.
Acronym: VEGENAT MED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Vegenat, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HULP 4985
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2019-02

CONDITIONS: Deglutition Disorders; Nutritional Deficiency; Chew Problems; Swallowing Disorder
Keywords: Deglutition disorders; Nutritional deficiency; Chew problems; Swallowing disorder; Nutritional formula; Nutritional oral supplement
MeSH Terms: conditions — Deglutition Disorders; Malnutrition | interventions — Control Groups; Educational Status; Guidelines as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Nutritional education, guidelines for the consumption of a completed shreded diet and recommendations for physical activity.
  Interventions: Other: Control Group (education, guidelines, recommendations)
- Experimental Group (Experimental): Nutritional education and guidelines for the consumption of a completed shreded diet including: 2 packets of 90 grams every day (One salted packet for lunch/dinner and one sweet packet for breakfast/afternoon snack) and recommendations for physical activity for one month.
  Interventions: Other: Experimental Group (education, guidelines, 2 pckts diet, recommendations)

INTERVENTIONS:
Other: Control Group (education, guidelines, recommendations) — Nutritional education and guidelines for the consumption of a completed shreded diet and recommendations for physical activity for one month.
  Arms: Control Group
Other: Experimental Group (education, guidelines, 2 pckts diet, recommendations) — Nutritional education and guidelines for the consumption of a completed shreded diet including 2 packets of 90 grams every day and recommendations for physical activity for one month.
  Arms: Experimental Group

SUMMARY:
Effect of a nutritional formula on the nutritional requirements in patients with chewing/swallowing problems during one month

DETAILED DESCRIPTION:
30 patients will receive nutritional education and guidelines for the consumption of a completed shreded diet including 2 packets of 90 grams every day (One salted packet for lunch/dinner and one sweet packet for breakfast/afternoon snack) and recommendations for physical activity for one month.

30 patients will receive nutritional education, guidelines for the consumption of a completed shreded diet and recommendations for physical activity during one month.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Individuals with chewing/swallowing disorder.
* Individuals well nourished or at malnutrition risk.
* Adequate cultural level and understanding of the clinical trial.
* Signed informed consent.

Exclusion Criteria:

* Individuals with body mass index ≥40 kg/m2.
* Individuals with acute, severe or chronic disease without control.
* Individuals with major surgeries during the last month.
* Individuals with gastrointestinal surgery the last three months.
* Individuals with moderate/severe cognitive impairment.
* Individuals with severe malnutrition.
* Individuals with amyotrophic lateral sclerosis.
* Individuals who consume nutritional oral supplements seven days prior to the start of the study.
* Enteral or parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of nutritional changes with regard to the nutritional requirements recommended | Up to one month
  Change percentage = (energy consumption at the end of the intervention period - energy consumption at the beginning of the intervention period) / energy consumption at the beginning of the intervention period * 100

SECONDARY OUTCOMES:
Change from Baseline Anthropometric Parameters | Up to one month
  Weight and Height to calcule BMI in kg/m2
Change from Baseline Anthropometric Parameters | Up to one month
  Waist Circumference
24h Dietary Recall Questionnaire | Up to one month
  Food and activity habits of people
Adverse Effects | Up to one month
  Gastrointestinal Symptoms (Nausea, Diarrhea, Bloating and other disorders)
Sensory perception | Up to one month
  Sensory Perception Scale
Functionality Variables | Up to one month
  Force dynamometry hand
Tolerance and adverse effects | Up to one month
  Tolerance and adverse effects questionnaire
International Physical Activity Questionnaire | Up to one month
  Activity habits of people

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, PhD, MS, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided